CLINICAL TRIAL: NCT01704157
Title: A Prospective Non-Randomized Unblinded Study Evaluating the Treatment of Knee Osteoarthritis With the Cryo-Touch III Device
Brief Title: A Prospective Study Evaluating the Treatment of Knee Osteoarthritis With the Cryo-Touch III Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MYO-0601; Pain-OA (Other: MyoScience)
Record Dates: First submitted 2012-10-05; First posted 2012-10-11 (Estimated); Results first posted 2023-09-29 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; knee; chronic pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Treatment (Other): Treatment with Cryo-Touch III Device
  Interventions: Device: Cryo-Touch III

INTERVENTIONS:
Device: Cryo-Touch III — Study treatment at Day 0.

SUMMARY:
A proof of concept study to evaluate the feasibility of safe and effective treatment through optimization of the Cryo-Touch III device for temporary relief of pain.

DETAILED DESCRIPTION:
Over 100 million patients in the United States suffer from chronic pain. Chronic pain conditions are often debilitating, taking a toll on a patient's physical and mental welfare. Though a variety of pain management techniques currently exist, the most common nonsurgical options provide slow-acting and/or short-term relief. Medication, often in the form of non-steroidal anti-inflammatory drugs (NSAIDs) and opioids, comes with an array of side effects such as nausea and vomiting. Medication also presents the possibility of more serious effects such as increased risk of heart attack and stroke, and tolerance or dependency issues. Surgical strategies tend to be reserved for more severe cases and are limited by the risks and complications typically associated with surgery including bleeding, bruising, scarring, and infection. A nonsurgical, minimally invasive, long-lasting approach to chronic pain management is desirable.

The Cryo-Touch III is a pain management device developed for a novel, minimally invasive procedure using focused cold therapy to target sensory nerve tissue and offer long-lasting pain relief through cryoanalgesia. The device operates on the well-established cryobiology principle that localized exposure to controlled moderately low temperature conditions can alter tissue function. The therapy treats nerves with low temperatures via a cold probe in the form of an assembly of small diameter needles, creating a highly localized treatment zone around the probe. This focused cold therapy creates a conduction block that prevents nerve signaling.

Though studies have proven efficacious in targeting motor nerves, the device's effect on sensory nerves has yet to have been investigated in the clinical setting. The goal of the study described herein is to evaluate the degree and duration of effect of the Cryo-Touch III in reducing chronic pain by targeting sensory nerves.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age and older.
* Participants must meet American College of Rheumatology (ACR) criteria for osteoarthritis of the knee (unilateral or bilateral). Clinical criteria includes knee pain and at least three of the following 6 criteria: 50 years of age or older, stiffness lasting less than 30 minutes, crepitus, bony tenderness, bony enlargement, and/or no warmth to the touch.
* Any medications (prescription and/or over-the counter) must be maintained on a stable schedule for ≥ 2 weeks prior to treatment. No washout period is allowed.
* An average Visual Analog Scale (VAS) for pain ≥ 4 over the last 30 days.
* Subject is willing and able to give written informed consent.
* Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
* Subject is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* A partial or full knee replacement (in the treated knee).
* Any use of systemic injections (in any area) within the last 6 months.
* Current enrollment in an investigational drug or a device study that specifically targets pain treatment.
* Any additional diagnosis that in the opinion of the investigator may directly contribute to knee pain.
* Any concomitant inflammatory disease or other condition that affects the joints (e.g. rheumatoid arthritis, metabolic bones disease, gout, active infection, etc.).
* Any clotting disorder and/or has used an anticoagulant (e.g., warfarin, clopidogrel, etc.) within seven (7) days prior to administration of the device.
* Allergy or intolerance to lidocaine.
* Any local skin condition at the treatment site that in the investigator's opinion would adversely affect treatment or outcomes.
* Any chronic medical condition that in the investigator's opinion would prevent adequate participation.
* Any chronic medication use (prescription, over-the-counter, etc.) that in the investigator's opinion would affect study participation or subject safety.
* For any reason, in the opinion of the investigator, the subject may not be a suitable candidate for study participation (i.e., history of noncompliance, drug dependency, any related knee injury due to a worker's compensation claim, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Neurovations, Napa, California
  - Injury Care Medical Center, Boise, Idaho

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were prospectively enrolled at 2 sites. Enrollment was initiated September 18, 2012 and completed March 25, 2013.
Period: Overall Study
Arm/Group | Open Treatment
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Treatment: Cryo-Touch III Device
Arm/Group | Open Treatment
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 12
  Gender: Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 33
Average Baseline Pain Score- Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — Visual Analog Scale, 0-10 where a higher score indicates greater intensity
  units on a scale | 6.3 (1.6)
Average Baseline Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale [Mean (Standard Deviation); unit: units on a scale] — The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale.
  A tri-dimensional, disease-specific, patient-reported outcome measure. Consists of 24 questions: 5 pain, 2 stiffness and 17 function. Each category contains a set of questions rated by the Subject on a 0-10 scale;
  The highest possible score was 50 for pain, 20 for stiffness and 170 for function, based on the 0-10 scale used to assess each question.
  The total score range is 0 to 240 with higher scores correlating to worse outcomes.
  units on a scale | 125.8 (42.8)

OUTCOME MEASURES:

1. Primary Outcome: Average Improvement in VAS Pain Score From Baseline to Day 7
Description: Visual Analog Scale(VAS), where a higher score indicates greater intensity; 0= no pain, 10=worst pain
Time Frame: Baseline to Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Treatment
Number analyzed (Participants) | 33
score on a scale | 2.2 (2.2)

2. Primary Outcome: Improvement in WOMAC Index From Baseline to Day 7
Description: The Western Ontario and McMaster Universities Osteoarthritis (WOMAC) pain scale.
  A tri-dimensional, disease-specific, patient-reported outcome measure. Consists of 24 questions: 5 pain, 2 stiffness and 17 function. Each category contains a set of questions rated by the Subject on a 0-10 scale;
  The highest possible score was 50 for pain, 20 for stiffness and 170 for function, based on the 0-10 scale used to assess each question.
  The total score range is 0 to 240 with higher scores correlating to worse outcomes.
Time Frame: Baseline to Day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Treatment
Number analyzed (Participants) | 33
score on a scale | 85.7 (53.4)

3. Secondary Outcome: Number of Participants Who Experienced Continued Treatment Effect at Each Time Point
Description: Subjects were asked to report whether they experienced continued treatment effect at the timepoints indicated.
Time Frame: Visit 3 (Day 7), Visit 4 (Day 30), Visit 5 (Day 56)
Measure: Count of Participants; unit: Participants
Arm/Group | Open Treatment
Number analyzed (Participants) | 33
Participants
  Day 7 | 31
  Day 30 | 28
  Day 56 | 23

ADVERSE EVENTS:
Time Frame: Adverse events were collected from treatment day through Day 140
Arm/Group | Open Treatment
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33
Other Adverse Events (participants affected / at risk) | 9/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Treatment (N=33)
Tuberculosis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Treatment (N=33)
Right leg numbness (Nervous system disorders) | 1 (1)
nausea duringprocedure (Injury, poisoning and procedural complications) | 1 (1)
Seasonal Cold (Infections and infestations) | 1 (1)
Arm Laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Tenderness to palpation in thigh (Musculoskeletal and connective tissue disorders) | 1 (1)
clicking sound in knee with standing (Musculoskeletal and connective tissue disorders) | 1 (1)
tingling/pain in feet (Nervous system disorders) | 1 (1)
Left Leg numbness (Nervous system disorders) | 1 (1)
Pain/loss of full range of motion with pivot (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol (2013-06-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT01704157/Prot_000.pdf